CLINICAL TRIAL: NCT06236438
Title: A Randomized, Phase 2/3 Study to Evaluate the Optimal Dose, Safety, and Efficacy of Livmoniplimab in Combination With Budigalimab Plus Chemotherapy Versus Pembrolizumab Plus Chemotherapy in Untreated Metastatic Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study to Evaluate Adverse Events, Optimal Dose, and Change in Disease Activity, With Livmoniplimab in Combination With Budigalimab Plus Chemotherapy Versus IV Infused Pembrolizumab Plus Chemotherapy in Adult Participants With Untreated Metastatic Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Acronym: LIVIGNO-4
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-721; 2023-505773-32-00 (Other: EU CT)
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Untreated Metastatic Non-Squamous Non-Small Cell Lung Cancer; NSCLC; Livmoniplimab; Budigalimab; Pembrolizumab; Chemotherapy; ABBV-181; ABBV-151
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — budigalimab; pembrolizumab; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Stage 1 (Cohort 1): Livmoniplimab Dose A (Experimental): Participants will receive livmoniplimab (dose A)+ budigalimab, + chemotherapy for 4 cycles followed by livmoniplimab + budigalimab + pemetrexed.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Stage 1 (Cohort 2): Livmoniplimab Dose B (Experimental): Participants will receive livmoniplimab (dose B) + budigalimab, + chemotherapy for 4 cycles followed by livmoniplimab + budigalimab + pemetrexed.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Stage 1 (Cohort 3): Budigalimab (Experimental): Participants will receive budigalimab + chemotherapy for 4 cycles followed by budigalimab + pemetrexed.
  Interventions: Drug: Budigalimab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Stage 1 (Cohort 4): Pembrolizumab (Experimental): Participants will receive pembrolizumab + chemotherapy for 4 cycles followed by pembrolizumab + pemetrexed.
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Stage 2 (Arm 1): Livmoniplimab (Dose Optimized) (Experimental): Participants will receive livmoniplimab (dose optimized) + budigalimab + chemotherapy for 4 cycles followed by livmoniplimab + budigalimab + pemetrexed.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Stage 2 (Arm 2): Placebo (Experimental): Participants will receive placebo + pembrolizumab + chemotherapy for 4 cycles followed by pembrolizumab + pemetrexed.
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Livmoniplimab — Intravenously (IV) Infusion
  Other Names: ABBV-151
  Arms: Stage 1 (Cohort 1): Livmoniplimab Dose A; Stage 1 (Cohort 2): Livmoniplimab Dose B; Stage 2 (Arm 1): Livmoniplimab (Dose Optimized)
Drug: Budigalimab — IV Infusion
  Other Names: ABBV-181
  Arms: Stage 1 (Cohort 1): Livmoniplimab Dose A; Stage 1 (Cohort 2): Livmoniplimab Dose B; Stage 1 (Cohort 3): Budigalimab; Stage 2 (Arm 1): Livmoniplimab (Dose Optimized)
Drug: Pembrolizumab — IV Infusion
  Arms: Stage 1 (Cohort 4): Pembrolizumab; Stage 2 (Arm 2): Placebo
Drug: Pemetrexed — IV Infusion
Drug: Cisplatin — IV Infusion
Drug: Carboplatin — IV Injection
Drug: Carboplatin — IV Infusion

SUMMARY:
Non-Squamous Non-Small Cell Lung Cancer (NSCLC) remains a leading cause of cancer mortality worldwide, with poor survival prospects for metastatic disease. The purpose of this study is to evaluate the optimized dose, adverse events, and efficacy of livmoniplimab in combination with budigalimab plus chemotherapy versus pembrolizumab plus chemotherapy in participants with untreated metastatic non-squamous non-small cell lung cancer.

Livmoniplimab is an investigational drug being developed for the treatment of NSCLC. There are 2 stages to this study. In Stage 1, there are 4 treatment arms. Participants will either receive livmoniplimab (at different doses) in combination with budigalimab (another investigational drug) + chemotherapy, budigalimab +chemotherapy, or pembrolizumab +chemotherapy. In Stage 2, there are 2 treatments arms. Participants will either receive livmoniplimab (optimized dose) in combination with budigalimab +chemotherapy or placebo in combination with pembrolizumab +chemotherapy. Chemotherapy consists of IV Infused pemetrexed + IV infused cisplatin or IV infused or injected carboplatin. Approximately 840 adult participants will be enrolled in the study across 200 sites worldwide.

Stage 1: In cohort 1, participants will receive intravenously (IV) infused livmoniplimab (dose A)+ IV infused budigalimab, + chemotherapy for 4 cycles followed by livmoniplimab + budigalimab + IV Infused pemetrexed. In cohort 2, participants will receive livmoniplimab (dose B) + budigalimab + chemotherapy for 4 cycles followed by livmoniplimab + budigalimab + pemetrexed. In cohort 3, participants will receive budigalimab + chemotherapy for 4 cycles followed by budigalimab + pemetrexed . In cohort 4, participants will receive IV Infused pembrolizumab + chemotherapy for 4 cycles followed by pembrolizumab + pemetrexed. Stage 2: In arm 1, participants will receive livmoniplimab (dose optimized) + budigalimab + chemotherapy for 4 cycles followed by livmoniplimab + budigalimab + pemetrexed. In arm 2, participants will receive IV Infused placebo + pembrolizumab + chemotherapy for 4 cycles followed by pembrolizumab + pemetrexed. The estimated study duration is 55 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, questionnaires, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically confirmed metastatic nonsquamous non-small cell lung cancer (NSCLC) with no known epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK) mutation, or other genomic aberration for which a locally approved targeted therapy is available.
* Must have at least 1 measurable lesion per response evaluation criteria in solid tumors (RECIST) v1.1 as determined by the local site Investigator/radiology assessment.
* Life expectancy of at least 3 months and adequate organ function.

Exclusion Criteria:

- Received prior systemic therapy for the treatment of metastatic NSCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Best Overall Response (BOR) of Complete Response (CR)/Partial Response (PR) | Up to 21 Months
  BOR of CR/PR is defined as achieving CR or PR according to response evaluation criteria in solid tumors (RECIST) v1.1 as determined by investigators at any time prior to subsequent anticancer therapy. Objective response rate (ORR), defined as the percentage of participants with a BOR of CR/PR, will be summarized.
Stage 2: Overall Survival (OS) | Up to 55 Months
  OS is defined as the time measured from randomization until death from any cause.

SECONDARY OUTCOMES:
Stage 1: Progression Free Survival (PFS) | Up to 21 Months
  PFS is defined as the time measured from randomization until the first documentation of progressive disease (PD) according to RECIST 1.1 as determined by investigators or death from any cause, whichever occurs first.
Stage 1: Duration of Response (DOR) | Up to 21 Months
  DOR is defined as the time from first CR/PR until the first documentation of PD according to RECIST 1.1 as determined by investigators or death from any cause, whichever occurs first.
Stage 1: OS | Up to 21 Months
  OS is defined as the time measured from randomization until death from any cause.
Stage 2: PFS | Up to 55 Months
  PFS is defined as the time measured from randomization until the first documentation of progressive disease according to RECIST 1.1 as determined by blinded independent central review (BICR) or death from any cause, whichever occurs first.
Stage 2: BOR of CR/PR | Up to 55 Months
  BOR of CR/PR is defined as achieving CR or PR according to RECIST 1.1 as determined by investigators at any time prior to subsequent anticancer therapy. ORR, defined as the percentage of participants with a BOR of CR/PR, will be summarized.
Stage 2: Change from Baseline in Physical Functioning (PF) as measured by the PF domain of European Organization for Research Treatment of Cancer Quality of Life Questionnaire 17 (EORTC QLQ-F17) | Up to 55 Months
  The EORTC QLQ-F17, a shorter, 17-item version that includes only the functional scales and the Global Health Status / Quality of Life scale of the EORTC QLQ-C30. QLQ-F17 includes the Physical (PF), Role (RF), Emotional (EF), Cognitive (CF) and Social Functioning (SF) scales as well as the Global Health Status/Quality of Life (QL) scale in their original wording. Participants rate items on a 4 point scale ranging form 1 to 4 (1- Not at All, 2= A Little, 3 = Quite a Bit, and 4= Very Much).
Stage 2: Change from Baseline in Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) | Up to 55 Months
  The NSCLC -SAQ scale with seven items assessing 5 symptoms of NSCLC (cough, pain, dyspnea, fatigue and poor appetites). The recall period is "over the last 7 days." Each item has a 5-point verbal rating scale from either 0 "No <symptom> at All" to 4 "Very severe <symptom>" or from 0 "Never" to 4 "Always," depending on the item's format.
Stage 2: Change from Baseline in Quality of Life as Measured by the Global Health Status/Quality of Life Domain of the EORTC QLQ-F17 | Up to 55 Months
  The EORTC QLQ-F17, a shorter, 17-item version that includes only the functional scales and the Global Health Status / Quality of Life scale of the EORTC QLQ-C30. QLQ-F17 includes the Physical (PF), Role (RF), Emotional (EF), Cognitive (CF) and Social Functioning (SF) scales as well as the Global Health Status/Quality of Life (QL) scale in their original wording. Participants rate items on a 4 point scale ranging form 1 to 4 (1- Not at All, 2= A Little, 3 = Quite a Bit, and 4= Very Much).
Stage 2: PFS per Investigator | Up to 55 Months
  PFS is defined as the time measured from randomization until the first documentation of progressive disease according to RECIST 1.1 as determined by the investigator or death from any cause, whichever occurs first.
Stage 1: BOR of CR/PR per Investigator | Up to 21 Months
  BOR of CR/PR is defined as achieving CR or PR according to RECIST 1.1 as determined by investigators. ORR, defined as the percentage of participants with a BOR of CR/PR, will be summarized.
Stage 2: DOR | Up to 55 Months
  DOR is defined as the time from first CR/PR until the first documentation of PD according to RECIST 1.1 as determined by BICR or death from any cause, whichever occurs first.
Stage 2: DOR per investigator | Up to 55 Months
  DOR is defined as the time from first CR/PR until the first documentation of PD according to RECIST 1.1 as determined by investigators or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (61):
- United States (19):
  - Moores Cancer Center /ID# 267782, La Jolla, California
  - Memorial Hospital West /ID# 262221, Pembroke Pines, Florida
  - Bond Clinic /ID# 262611, Winter Haven, Florida
  - University Cancer & Blood Cent /ID# 261824, Athens, Georgia
  - The University of Chicago Medical Center /ID# 262259, Chicago, Illinois
  - University of Kansas Medical Center /ID# 263196, Westwood, Kansas
  - Baptist Health Lexington /ID# 261823, Lexington, Kentucky
  - Cancer & Hematology Centers of Western Michigan - East /ID# 261826, Grand Rapids, Michigan
  - Washington University-School of Medicine /ID# 262759, St Louis, Missouri
  - Stony Brook Cancer Center /ID# 261954, Stony Brook, New York
  - Cone Health Cancer Center /ID# 262583, Greensboro, North Carolina
  - Oncology Hematology Care, Inc - Blue Ash /ID# 262733, Cincinnati, Ohio
  - Guthrie Robert Packer Hospital /ID# 262758, Sayre, Pennsylvania
  - Renovatio clinical /ID# 262000, El Paso, Texas
  - Houston Methodist Hospital /ID# 262722, Houston, Texas
  - Texas Oncology - Plano East /ID# 264356, Plano, Texas
  - Texas Oncology - San Antonio Medical Center - Research Drive /ID# 264311, San Antonio, Texas
  - Renovatio Clinical /ID# 261999, The Woodlands, Texas
  - Vista Oncology - East Olympia /ID# 262303, Olympia, Washington
- Australia (3):
  - Canberra Hospital /ID# 261891, Garran, Australian Capital Territory
  - Nepean Hospital /ID# 262157, Kingswood, New South Wales
  - Westmead Hospital /ID# 261894, Westmead, New South Wales
- Belgium (6):
  - Universitair Ziekenhuis Antwerpen /ID# 261270, Edegem, Antwerpen
  - Cliniques Universitaires UCL Saint-Luc /ID# 261267, Brussels, Brussels Capital
  - Hospital La Louviere Site Jolimont - Helora /ID# 261269, La Louvière, Hainaut
  - Groupe Sante CHC - Clinique du MontLegia /ID# 262338, Liège, Liege
  - AZ Maria Middelares /ID# 262313, Ghent
  - UCL Namur University Hospital, Site Sainte-Elisabeth /ID# 262557, Namur
- Chile (5):
  - Oncored /Id# 261801, Vitacura, Region Metropolitana Santiago
  - Centro de Investigacion y Desarrollo Oncologico /ID# 261800, Temuco, Región de la Araucanía
  - Sociedad Cem-Cancer Spa /Id# 262316, Viña del Mar, Región de Valparaíso
  - Fundacion Arturo Lopez Perez /ID# 261700, Providencia, Santiago Metropolitan
  - Hospital Clinico Universidad De Los Andes /ID# 262665, Santiago
- France (5):
  - APHM - Hopital Nord /ID# 261129, Marseille, Bouches-du-Rhone
  - CHU Grenoble - Hopital Michallon /ID# 261131, La Tronche, Isere
  - Institut Curie /ID# 261127, Paris, Paris
  - Hospices Civils de Lyon (HCL) - Hopital Louis Pradel /ID# 261644, Bron, Rhone
  - Centre Hosp Intercommunal de Creteil /ID# 261130, Créteil, Val-de-Marne
- Israel (2):
  - Shaare Zedek Medical Center /ID# 262432, Jerusalem, Jerusalem
  - Rambam Health Care Campus /ID# 262431, Haifa
- Japan (3):
  - National Cancer Center Hospital East /ID# 261923, Kashiwa-shi, Chiba
  - Saitama Prefectural Cancer Center /ID# 262703, Kitaadachi-gun, Saitama
  - National Cancer Center Hospital /ID# 261925, Chuo-ku, Tokyo
- Netherlands (3):
  - Ziekenhuis St. Jansdal /ID# 261193, Harderwijk, Gelderland
  - Zuyderland Medisch Centrum /ID# 261190, Heerlen, Limburg
  - Isala /ID# 262458, Zwolle, Overijssel
- Pan American Center for Oncology Trials /ID# 269666, Rio Piedras, Puerto Rico
- Spain (7):
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 262723, Santiago de Compostela, A Coruna
  - Institut Català d'Oncologia (ICO) - L'Hospitalet /ID# 262118, L'Hospitalet de Llobregat, Barcelona
  - UOMi Cancer Center - Clinica Tres Torres /ID# 262116, Barcelona
  - Hospital Universitario Vall de Hebron /ID# 262113, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 262114, Madrid
  - Hospital Universitario 12 de Octubre /ID# 262112, Madrid
  - Hospital Clinico Universitario de Valencia /ID# 262115, Valencia
- Taiwan (4):
  - National Cheng Kung University Hospital /ID# 262016, Tainan
  - Mackay Memorial Hospital /ID# 262534, Taipei
  - Taipei Medical University Hospital /ID# 262020, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 262535, Taoyuan
- Turkey (Türkiye) (3):
  - Gazi University Medical Faculty /ID# 261786, Ankara
  - Ankara City Hospital /ID# 261785, Ankara
  - Dr. Suat Seren Gogus Has /ID# 261789, Izmir

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-721